CLINICAL TRIAL: NCT00976755
Title: Everolimus First-line Therapy in Non-rapidly Progressive Castration Resistant Prostate Cancer (CRPC). A Multicenter Phase II Trial.
Brief Title: Everolimus as First-Line Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 08/08; SWS-SAKK-08/08; EU-20967; CDR0000649049
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; hormone-resistant prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A: Everolimus (Experimental): Everolimus:
  10mg daily
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — Everolimus:
  10mg daily
  Other Names: Afinitor®; Votubia®; RAD001

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying the side effects of everolimus and to see how well it works as first-line therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival at 12 weeks of patients with non-rapidly progressive castration-resistant prostate cancer treated with everolimus as first-line therapy.
* Assess the activity and safety of this regimen in these patients.

Secondary

* Determine the progression-free survival at 24 weeks of patients treated with this regimen.
* Determine the percentage of PSA response from baseline to 12 weeks in patients treated with this regimen.
* Determine the changes in PSA-doubling time in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up at 28 days and then every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or locally advanced adenocarcinoma of the prostate

  * No curative therapy available
  * Oligosymptomatic or asymptomatic patients
* Tumor progression after ≥ 1 hormonal treatment (orchiectomy or luteinizing-hormone releasing-hormone [LHRH] agonist) with documented total testosterone levels ≤ 1.7 nmol/L (≤ 50 ng/dL)

  * Concurrent LHRH agonist therapy is required for patients who have not been surgically castrated
  * Must have stopped antiandrogen therapy ≥ 6 weeks before the start of trial treatment without withdrawal response
* PSA progression defined as an increase in PSA ≥ 25% (and an absolute increase of 2 ng/mL or more) over nadir value on hormonal therapy measured on 3 successive occasions ≥ 1 week apart

  * If the third measurement is not higher than the second, a fourth measurement will be taken (patient allowed if the fourth measurement is higher than the second)
  * PSA doubling time ≥ 55 days
* No known or suspected CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 90 g/L
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Creatinine clearance ≥ 40 mL/min
* Fasting serum cholesterol ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 times ULN

  * Appropriate lipid-lowering medication allowed in case one or both of these thresholds are exceeded
* Patient compliance and geographic proximity that would allow proper staging and follow-up are required
* No malignancy within the past 5 years except curatively treated localized nonmelanoma skin cancer or Ta and Tis bladder cancer
* No known history of HIV
* No serologically confirmed hepatitis B or C
* No serious underlying medical condition that, in the judgment of the investigator, could impair the ability of the patient to participate in the trial including, but not limited to, any of the following conditions:

  * Uncontrolled or acute severe infection
  * Uncontrolled diabetes
  * Advanced chronic obstructive pulmonary disease
* No psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent, or interfering with compliance for oral drug intake
* No known hypersensitivity to trial drug or hypersensitivity to any of its components

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, radioisotopes, small molecules, immunotherapy, or investigational drug therapy for prostate cancer
* No local radiotherapy within the past 2 weeks
* No major surgery within the past 4 weeks
* No concurrent radiotherapy
* No concurrent angiotensin converting enzyme inhibitors
* No concurrent chronic immunosuppressive therapy including high-dose corticosteroids (i.e., > 25 mg prednisone equivalent per day)
* No products known to affect PSA levels (e.g., PC Calm, PC Plus, PC SPES, finasteride, or fluconazole) within the past 4 weeks or concurrently
* No strong CYP3A4 inhibitors (e.g., itraconazole, erythromycin, clarithromycin, diltiazem, verapamil, or grapefruit or its juice) within the past 2 weeks or concurrently
* No strong CYP3A4 inducers (e.g., phenytoin, rifampicin, carbamazepine, phenobarbital, or St. John wort) within the past 2 weeks or concurrently
* No concurrent bisphosphonates

  * Patients must continue to receive bisphosphonates regularly if it was started prior to entering the trial
* No concurrent experimental drugs or other anticancer therapy in a clinical trial within the past 30 days
* No concomitant drugs contraindicated for use with the trial drug according to the investigator's drug brochure

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2012-11-29 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 12 weeks | at 12 weeks
  PFS at 12 weeks is defined as the absence of disease progression or death at 12 weeks after start of treatment.

SECONDARY OUTCOMES:
PFS at 24 weeks | at 24 weeks
  PFS at 24 weeks is defined as the absence of any disease progression or death at 24 weeks after start of treatment.
Progression-free survival | from start of treatment until progression or death of any cause
  from start of treatment until progression or death of any cause, whereas it will be censored at the last follow-up visit or initiation of a different treatment.
Adverse events (AEs) according to NCI CTCAE v. 3.0 | from start of treatment until progression or death of any cause
  All AEs will be assessed according to NCI CTCAE v3.0
PSA response | 50% and 30%, best and at 12 weeks
  50% PSA response is defined as a decrease in PSA level of at least 50% (compared to baseline PSA).
  30% PSA response is defined as a decrease in PSA level of at least 30% (compared to baseline PSA).
  Best response is defined as the percentage of change in PSA from baseline to the maximum decline in PSA at any point under treatment.
  Response at 12 weeks is defined as the percentage of change in PSA from baseline to 12 weeks (or earlier for those patients who discontinue therapy, in this case last PSA values recorded should be taken).
Changes in PSA-doubling time | Time points for later calculations include: after 12 weeks, after 24 weeks and at best PSA response
  PSA-DT is calculated by natural log of 2 divided by the slope of the relationship between the log of PSA and time of PSA measurement for each patient.
Tumor assessment of measurable disease according to RECIST v1.1 criteria | The first assessment will be performed after 12 weeks of treatment, or earlier if clinically indicated.
  For patients with measurable disease at baseline RECIST v1.1 will be used to define CR, PR, SD and PD.
Tumor assessment of bone lesions | at 12 weeks.
  Bone metastases can be assessed by radionuclide bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: Arnoud Templeton, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Silke Gillessen, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (12):
- Switzerland (12):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Templeton A, Rothermundt C, Cathomas R, et al.: Everolimus as first-line therapy in nonrapidly progressive metastatic castration-resistant prostate cancer (mCRPC): A multicenter phase II trial (SAKK 08/08). [Abstract] J Clin Oncol 29 (Suppl 15): A-4588, 2011.
- [Derived] Templeton AJ, Dutoit V, Cathomas R, Rothermundt C, Bartschi D, Droge C, Gautschi O, Borner M, Fechter E, Stenner F, Winterhalder R, Muller B, Schiess R, Wild PJ, Ruschoff JH, Thalmann G, Dietrich PY, Aebersold R, Klingbiel D, Gillessen S; Swiss Group for Clinical Cancer Research (SAKK). Phase 2 trial of single-agent everolimus in chemotherapy-naive patients with castration-resistant prostate cancer (SAKK 08/08). Eur Urol. 2013 Jul;64(1):150-8. doi: 10.1016/j.eururo.2013.03.040. Epub 2013 Apr 6. PMID 23582881